CLINICAL TRIAL: NCT00336128
Title: Population Based Intervention to Prevent Obesity in Kindergartens (TigerKids)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Child Health Foundation (Other); Bavarian State Ministry of Environment, Public Health and Consumer Protection (Other Government); Bavarian Health and Food Safety Authority (LGL) (Unknown); Institute for Social Paediatrics and Adolescent Medicine, Munich (Unknown); State Institute of Early Childhood Research, Munich (Unknown); AOK.Die Gesundheitskasse (Industry); Research Centre for Physical Education and Sports of Children and Adolescents, Karlsruhe (Unknown)
Responsible Party: Principal Investigator, Prof. Berthold Koletzko, Prof. Dr., Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UGV 03050904006
Record Dates: First submitted 2006-06-12; First posted 2006-06-13 (Estimated); Last update posted 2022-04-13 (Actual); Status verified 2020-09

CONDITIONS: Obesity
Keywords: infant; kindergarten; obesity; adiposity
MeSH Terms: conditions — Obesity

INTERVENTIONS:
Behavioral: attitude change — TigerKids: setting based prevention program to reduce obesity risk factors in children
Behavioral: adiposity prevention program — The behavioral intervention aimed at modifying physical activity and food and drink choices at the kindergarten setting

SUMMARY:
Behavioral intervention at Kindergarten setting aiming at increased fruit and vegetable consumption, decreased intake of high energy foods, snacks, sweets, increased intake of water/low energy drinks, decreased intake of high energy drinks. Physical activity should be more than 1 hour/day and TV/media consumption less than 1 hour/day.

Main questions are:

Do children differ in intervention and control kindergartens according to their nutrition behaviour? Do children in the intervention kindergartens have a higher physical training than such in the control kindergartens? Data were collected with a standardised questionnaire.

Do children differ in intervention and control kindergartens according to their body mass index?

DETAILED DESCRIPTION:
The program is based on actual cognitions and methods of the early education science. In the initial phase study part I (2003-2006) we will study over three years in 75 kindergartens of four administrative districts in Bavaria, Germany: Bamberg, Günzburg, Ingolstadt and Schwandorf.

The objective of the study part II is to evaluate the effects of the TigerKids intervention program on overweight prevalence in childhood. Data concerning BMI, nutrition behavior and physical activity are assessed both at baseline (September/October 2007) and after 10 months intervention in > 450 control- and intervention-kindergartens in Bavaria.

ELIGIBILITY:
Inclusion Criteria:

* infant of intervention- or control-kindergarten

Exclusion Criteria:

* absence of parenteral consent to participate

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30000 (Estimated)
Dates: Start 2003-10; Primary Completion 2006-05 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Body mass index | 2005, 2006, 2007, 2008
nutrition behavior | 2005, 2006, 2007, 2008
physical activity | 2005, 2006, 2007, 2008

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Koletzko, Prof., Principal Investigator — Ludwig-Maximilians-Universitaet

REFERENCES:
- [Derived] Bayer O, von Kries R, Strauss A, Mitschek C, Toschke AM, Hose A, Koletzko BV. Short- and mid-term effects of a setting based prevention program to reduce obesity risk factors in children: a cluster-randomized trial. Clin Nutr. 2009 Apr;28(2):122-8. doi: 10.1016/j.clnu.2009.01.001. Epub 2009 Mar 20. PMID 19303675